CLINICAL TRIAL: NCT07190157
Title: Evaluation of the Relationship Between Ductus Venosus Doppler Parameters and Perinatal Outcomes in Pregnancies With and Without Intrauterine Growth Restriction
Brief Title: Relationship of DV Doppler Parameters to Perinatal Outcomes in IUGR vs Non-IUGR
Acronym: DV-FGR
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024/212
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fetal Growth Restriction; Perinatal Outcome; Pregnancy, High Risk
Keywords: Perinatal Outcome; Fetal Growth Restriction; Pregnancy
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IUGR Group: Pregnant women with singleton fetuses between 24-37 weeks of gestation, with abdominal circumference (AC) and/or estimated fetal weight (EFW) below the 10th percentile.
- Control Group: Pregnant women with singleton fetuses between 24-37 weeks of gestation, with AC and/or EFW between the 10th and 90th percentile (appropriate-for-gestational-age).

SUMMARY:
This observational study investigates whether blood flow in the ductus venosus, a small fetal vein measured by Doppler ultrasound, is related to pregnancy outcomes. A total of pregnant women with and without intrauterine growth restriction (IUGR) will be examined between 24 and 37 weeks of gestation. Ductus venosus Doppler parameters will be recorded and compared with perinatal outcomes such as Apgar scores, neonatal intensive care unit admission, and perinatal mortality. The aim of this research is to improve the early identification of high-risk pregnancies and to support better monitoring and management strategies for fetal health.

DETAILED DESCRIPTION:
Detailed Description:

Intrauterine growth restriction (IUGR) is a major cause of perinatal morbidity and mortality and has been associated with impaired fetal circulation. The ductus venosus (DV) plays a critical role in fetal hemodynamics by directing oxygenated blood to the heart and brain. Abnormal DV Doppler waveforms have been linked to adverse perinatal outcomes, particularly in growth-restricted fetuses.

This prospective observational case-control study will include approximately 160 singleton pregnancies between 24 and 37 weeks of gestation, of which 80 will be diagnosed with IUGR and 80 will be healthy controls. Doppler parameters of the DV, including pulsatility index, peak velocity, and a-wave characteristics, will be measured. These values will be correlated with perinatal outcomes such as Apgar scores, neonatal intensive care unit admission, and perinatal mortality.

The study is expected to provide further insight into the predictive value of DV Doppler in differentiating high-risk pregnancies and to contribute to improved prenatal surveillance and management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies between 24 and 37 weeks of gestation Singleton pregnancies with abdominal circumference (AC) and/or estimated fetal weight (EFW) below the 10th percentile for gestational age Singleton pregnancies with abdominal circumference (AC) and/or estimated fetal weight (EFW) between the 10th and 90th percentiles for gestational age

Exclusion Criteria:

Multiple pregnancies Pregnancies with major fetal structural anomalies or chromosomal abnormalities Pregnant women with maternal systemic comorbidities (e.g., diabetes mellitus, chronic hypertension, renal disease, autoimmune disorders) Pregnancies in women under 18 years of age Presence of perinatal infection Pregnancies conceived by in vitro fertilization (IVF)

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group/Cohort 1: IUGR Group Title: IUGR Group Description: Pregnant women with singleton fetuses between 24-37 weeks of gestation, with abdominal circumference (AC) and/or estimated fetal weight (EFW) below the 10th percentile.
  Group/Cohort 2: Control Group Title: Control Group Description: Pregnant women with singleton fetuses between 24-37 weeks of gestation, with AC and/or EFW between the 10th and 90th percentile (appropriate-for-gestational-age).
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Perinatal Mortality | From delivery up to 7 days postpartum
  Death of the fetus or neonate, including stillbirth and neonatal death.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gölbasi, Study Director — Izmir City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Izmir city hospital, Izmir, BAYRAKLI
  - Izmir City Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No
NO,

REFERENCES:
- [Background] Fratelli N, Amighetti S, Bhide A, Fichera A, Khalil A, Papageorghiou AT, Prefumo F, Thilaganathan B. Ductus venosus Doppler waveform pattern in fetuses with early growth restriction. Acta Obstet Gynecol Scand. 2020 May;99(5):608-614. doi: 10.1111/aogs.13782. Epub 2019 Dec 22. PMID 31784981
- [Background] Cruz-Martinez R, Figueras F, Benavides-Serralde A, Crispi F, Hernandez-Andrade E, Gratacos E. Sequence of changes in myocardial performance index in relation to aortic isthmus and ductus venosus Doppler in fetuses with early-onset intrauterine growth restriction. Ultrasound Obstet Gynecol. 2011 Aug;38(2):179-84. doi: 10.1002/uog.8903. Epub 2011 Jul 15. PMID 21154784